CLINICAL TRIAL: NCT01299077
Title: A Retrospective Drug Use Survey (DUS) of Triple Therapy (Methycobal (MBL)+ Myonal (MYO)+ Non-steroidal Anti-inflammatory Drags (NSAID)) on the Symptom Relief of Lumbar Disc Degenerative Disease in China
Brief Title: Drug Use Survey (DUS) of Triple Therapy (Methycobal (MBL)+ Myonal (MYO)+ Non-steroidal Anti-inflammatory Drags (NSAID)) on the Symptom Relief of Lumbar DDD in China
Status: Completed | Type: Observational
Sponsor: Eisai China Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: EISAI-MBL-2010-1
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2011-11-28 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2011-05

CONDITIONS: Lumbar Disc Degenerative Disease
Keywords: Lumbar disc degenerative disease; Methycobal
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lumbar disc degenerative disease: Triple therapy (MBL+ MYO+ NSAIDs) which prescribed by doctors (Drs) based on disease condition

SUMMARY:
The purpose of this study is to observe the overall satisfaction of patients with degenerative disc disease after receiving triple therapy.

DETAILED DESCRIPTION:
DDD (lumbar disc degenerative disease ) patients who have been prescribed triple therapy (MBL+ MYO+ NSAIDs) over 2 weeks of triple therapy were enrolled in the study. They were asked to assess their overall satisfaction degree on triple therapy.

ELIGIBILITY:
Inclusion criteria:

1. lumbar degenerative disc disease (DDD)
2. patients who have been prescribed over 2 weeks of triple therapy

Exclusion criteria:

Patients who do not meet inclusion criteria for DDD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients visited to the clinics with lumbar disc degenerative disease
Sampling Method: Non-Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Song, Study Director — Eisai China Inc.
Locations (10):
- China (10):
  - Dongfang Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shao Yifu Hospital of Zhejiang University, Hanzhou, Zhejiang
  - The 1st Hospital of Zhejiang University, Hanzhou, Zhejiang
  - The 1st People Hospital of Hanzhou, Hanzhou, Zhejiang
  - The 2nd Hospital of Zhejiang University, Hanzhou, Zhejiang
  - Traditional Chinese Medicine Hospital of Zhejiang, Hanzhou, Zhejiang

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 10 centers in China during the period of 09-Jun-2010 to 28-Sept-2010 .
Groups:
- Lumbar Disc Degenerative Disease: Triple therapy ( Methycobal (MBL) + Myonal (MYO) + non-steroidal anti-inflammatory drugs (NSAIDs)) which prescribed by doctors (Drs) based on disease condition. MBL 0.5 mg : three times daily for two weeks, MYO 50 mg : three times daily for two weeks:
  NSAID (diclofenac) 75 mg,: twice daily for two weeks
Period: Overall Study
Arm/Group | Lumbar Disc Degenerative Disease
Started | 478
Completed | 478
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lumbar Disc Degenerative Disease
Number analyzed (Participants) | 478
Age Continuous [Mean (Standard Deviation); unit: years] | 50.34 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252
  Male | 226
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 478
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Satisfaction Degree After 2 Weeks Treatment of Triple Therapy (MBL+MYO+NSAID).
Description: The measurement of overall satisfaction degree was in three scales, that was satisfactory, just so so and dissatisfactory. The measurement was estimated by both the physicians and the patients respectively.
Time Frame: 2 weeks
Population: The primary analysis will be on the Per-protocol (PP) population. PP population includes all subjects who received the dose of study drug without protocol deviation and had all the assessment per protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Lumbar Disc Degenerative Disease
Number analyzed (Participants) | 478
percentage of participants
  Estimation by Physicians: satisfactory | 91.21
  Estimation by Physicians: just so so | 7.74
  Estimation by Physicians: dissatisfactory | 1.05
  Estimation by Patients: satisfactory | 86.4
  Estimation by Patients: just so so | 12.76
  Estimation by Patients: dissatisfactory | 0.84

2. Secondary Outcome: Onset Time of Symptom Relief.
Description: Kaplan-Meier Estimates for the Average Onset Time of Symptom Relief. In this case the onset time of symptom relief was defined as the days between the end of triple therapy and the symptom improvement reported by patients.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Average Days of Onset Time
Arm/Group | Lumbar Disc Degenerative Disease
Number analyzed (Participants) | 478
Average Days of Onset Time | 4.68 (2.61)

3. Secondary Outcome: Safety Data During Triple Therapy.
Description: Percentage of participants with reported Adverse Events (AE) and Serious Adverse Event (SAE)
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Lumbar Disc Degenerative Disease
Number analyzed (Participants) | 478
Percentage of participants
  AE | 2.7
  SAE | 0

4. Secondary Outcome: Japanese Orthopedic Association (JOA) Score
Description: Each patient is Scored on JOA at baseline and two weeks. JOA is short for Japanese Orthopedic Association, which consists of 12 items: low back pain, lower extremity pain and numbness, walking ability, straight leg raising, muscle strength, sensory and etc. The first 3 item's scores are range from 0 to 3 and the others are from 0 to 2. Higher score means better condition.
  All of these items scores are combined for a total overall JOA score, which is range from 0 to 27.
Time Frame: Baseline and 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on JOA
Arm/Group | Lumbar Disc Degenerative Disease
Number analyzed (Participants) | 478
Scores on JOA
  Baseline | 15.72 (3.51)
  2 weeks | 21.28 (3.41)

5. Secondary Outcome: Visual Analogue Scale (VAS) Score
Description: Each patient is Scored on VAS at baseline and two weeks. VAS is the abbreviation of visual analogue score. There is no subscale in VAS. The maximum value of vas is 10 and the minimum is 0. This is self-evaluation method to present the severity of patient pain. More score number, more pain.
Time Frame: Baseline and 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on VAS
Arm/Group | Lumbar Disc Degenerative Disease
Number analyzed (Participants) | 478
Scores on VAS
  Baseline | 6.23 (1.38)
  2 weeks | 2.61 (1.70)

ADVERSE EVENTS:
Arm/Group | Lumbar Disc Degenerative Disease
Serious Adverse Events (participants affected / at risk) | 0/478
Other Adverse Events (participants affected / at risk) | 13/478
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumbar Disc Degenerative Disease (N=478)
Abdominal discomfort (Gastrointestinal disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No